CLINICAL TRIAL: NCT00076674
Title: Levetiracetam Treatment of L-dopa Induced Dyskinesias
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 040101; 04-N-0101
Record Dates: First submitted 2004-01-28; First posted 2004-01-29 (Estimated); Last update posted 2016-09-22 (Estimated); Status verified 2005-10

CONDITIONS: Dyskinesias; Parkinson Disease
Keywords: Parkinson's Disease; Keppra; Motor Fluctuations; Intravenous Levodopa; Antiparkinsonian Response; Parkinson Disease; PD
MeSH Terms: conditions — Dyskinesias; Parkinson Disease

INTERVENTIONS:
Drug: Intravenous Levodopa

SUMMARY:
This study will evaluate the effects of levetiracetam (Keppra (Trademark) on Parkinson's disease symptoms and on dyskinesias (involuntary movements) that develop as a result of long-term treatment with levodopa. Levetiracetam blocks certain protein receptors on brain cells and thus can change the spread of brain signals believed to be affected in patients with Parkinson's disease.

Patients between 30 and 80 years of age with relatively advanced Parkinson's disease and dyskinesias due to levodopa therapy may be eligible for this 6-week study.

Screening and baseline evaluation - Participants are evaluated with a medical history, physical examination and neurologic evaluation, blood tests, urinalysis, electrocardiogram (EKG), 24-hour holter monitor (heart monitoring), and cardiology consultation. A chest x-ray and MRI or CT scan of the brain are done if needed. If possible, patients stop taking all antiparkinsonian medications except levodopa (Sinemet) for one month (2 months if taking Selegiline) before the study begins and throughout its duration. (If necessary, patients may use short-acting agents, such as Mirapex, Requip or Amantadine.)

Dose-finding phase - Patients are admitted to the NIH Clinical Center for 2 to 3 days for a levodopa "dose-finding" procedure. For this test, patients stop taking Sinemet and instead have levodopa infused through a vein. During the infusions, the drug dose is increased slowly until parkinsonian symptoms improve or unacceptable side effects occur or the maximum study dose is reached. Symptoms are monitored frequently. (Patients who have had dosing infusions in the last 3 months do not have to undergo this phase of the study.)

Active study phase - Patients are randomly assigned to take levetiracetam or placebo ("sugar pill") twice a day for 6 weeks. At the end of weeks 1, 2 4, and 5, patients come to the clinic for blood tests, an EKG, and a review of adverse side effects. At the end of weeks 3 and 6, patients are hospitalized to study the response to treatment. They again stop taking Sinemet and selegiline and their ability to perform motor tasks is evaluated. They are then placed on an L-dopa infusion for 10 hours. Placebo may be infused at various times instead of L-dopa. Motor symptoms are evaluated several times during the infusion. Blood is drawn once during the infusion for research studies.

Lumbar puncture - Patients undergo a lumbar puncture (spinal tap) at the end of weeks 1 and 4 to measure certain brain chemicals and drug levels. For this test, a local anesthetic is given and a needle is inserted in the space between the vertebrae in the lower back. About 2 tablespoons of fluid is collected through the needle.

Magnetic resonance imaging (MRI) - Patients with changing disease activity may undergo MRIs at baseline, at the end of week 1 and at the end of the study to show changes in the brain. The patient lies in a narrow cylinder (the scanner) that uses radio waves and a magnetic field to produce images of the brain, which show structural and chemical changes.

Follow-up - 2 weeks after the study ends, patients are contacted by phone for a review of side effects or they return to the clinic for an evaluation.

DETAILED DESCRIPTION:
Introduction: Parkinson's disease is a progressive degenerative disease of unknown etiology. Its treatment has been symptomatic and the most successful approach has been to replace the missing dopamine through administration of its precursor levodopa. As the disease progresses the usefulness of this approach gradually diminishes and motor complications become a source of significant disability. Although a number of pharmacological strategies have attempted to improve this situation, none has yet proven fully satisfactory. The mechanism by which levetiracetam exerts this beneficial effect is unknown. Recently, in a PD monkey model levetiracetam was found to moderate dyskinesias and other motor complications, possibly due to its effects on striatal GABAergic transmission.

Objective: To evaluate the acute ability of levetiracetam to safely ameliorate dopaminomimetic-treatment-associated dyskinesias and related motor complications in parkinsonian patients without compromising the antiparkinsonian response.

Study Population: 22 moderately advanced parkinsonian patients will be enrolled into a randomized, placebo controlled, double-blind proof-of-principle study. Levetiracetam efficacy will be assessed through the use of validated motor function scales. Safety will be monitored by means of frequent clinical evaluations and laboratory tests.

Anticipated Risks and Benefits: The potential risks associated with this study amount to only a minor increase over minimal risk and are primarily associated with adverse reactions to the medications involved. Levetiracetam is a marketed drug with a wide margin of safety. Patients receiving drug could benefit from improvement of their symptoms, those on placebo will also have their medications adjusted, leading to an improved quality of life.

Outcome Estimate and Potential Meaning for the Field: This study should further the understanding of mechanisms contributing to motor disability in patients with PD that may lead to the development of improved therapeutic interventions for this disorder and for associated motor response complications.

ELIGIBILITY:
INCLUSION CRITERIA:

Patients who meet all of the following inclusion criteria will be able to participate in the study:

1. Patient is between the ages of 30 and 80, inclusive;
2. Patient has been diagnosed with idiopathic Parkinson's disease based on the presence of a characteristic clinical history and neurological findings;
3. Patient has relatively advanced disease with levodopa-associated motor response complications, including peak-dose dyskinesias and wearing-off fluctuations ;
4. Patient is willing to adhere to protocol requirements as evidenced by written, informed consent.

EXCLUSION CRITERIA:

Patients meeting any of the following exclusion criteria will not be enrolled or immediately withdrawn from the study, as appropriate:

1. Patient has a history of any medical condition that can reasonably be expected to subject them to unwaranted risk;
2. Patient has clinically significant laboratory abnormalities including impaired renal function (CL(cr) equals 30-50 ml/min.);
3. Patient is uable to br treated with levodopa/carbidopa alone or with a single, relatively short-acting dopamine agonist, such as pramipexole or ropinirole;
4. Patient is taking a prohibited concomitant medication;
5. Patient has not been using or was not continuing to use an adequate contraceptive method for the last 30 days, or is not at least one year post-menopausal (if female);
6. Patient is pregnant or breastfeeding;
7. Patient is implanted with bilateral deep brain stimulators;
8. Patient has prior pallidotomy or other ablative surgeries for treatment of PD;
9. Patient has cognitive impairment (MMSE less than 25);
10. Patient has participated in a clinical study with an investigational drug within the last 30 days;
11. Patient has a condition (such as active drug or alcohol abuse) that, in the opinion of the investigators, would interfere with compliance or safety;
12. Patient is unwilling to sign an informed consent or to comply with protocol requirements;
13. Patient has a history of psychiatric illness.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40
Dates: Start 2004-01; Study Completion 2005-10

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Neurological Disorders and Stroke (NINDS), Bethesda, Maryland, United States

REFERENCES:
- [Background] Bernheimer H, Birkmayer W, Hornykiewicz O, Jellinger K, Seitelberger F. Brain dopamine and the syndromes of Parkinson and Huntington. Clinical, morphological and neurochemical correlations. J Neurol Sci. 1973 Dec;20(4):415-55. doi: 10.1016/0022-510x(73)90175-5. No abstract available. PMID 4272516
- [Background] Kish SJ, Shannak K, Hornykiewicz O. Uneven pattern of dopamine loss in the striatum of patients with idiopathic Parkinson's disease. Pathophysiologic and clinical implications. N Engl J Med. 1988 Apr 7;318(14):876-80. doi: 10.1056/NEJM198804073181402. PMID 3352672
- [Background] Mizuno Y, Mori H, Kondo T. Parkinson's disease: from etiology to treatment. Intern Med. 1995 Nov;34(11):1045-54. doi: 10.2169/internalmedicine.34.1045. PMID 8774962